CLINICAL TRIAL: NCT02510482
Title: Biological Variation of Cardiac Biomarkers in Aortic Valve Stenosis
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 15-2-023
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2016-09

CONDITIONS: Aortic Valve Stenosis
Keywords: cardiac biomarkers
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Aortic valve stenosis: Individuals with clinically stable moderate aortic valve stenosis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Calcified aortic valve stenosis (CAVS) is a progressive disease and nowadays, the cornerstone in diagnostics and follow-up is echocardiography. Cardiac biomarkers (such as cardiac troponins T and I and NT-pro-BNP) hold promise to fulfil a role in early recognition of complications concerning the aortic valve and decompensation. For this purpose, it is important to assess the normal biological variation (BV) of cardiac biomarkers in CAVS. The assessment of biological variation will contribute to a better understanding of fluctuation of cardiac biomarkers in subjects with stable CAVS. These data will improve monitoring of CAVS using cardiac biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable moderate aortic valve stenosis
* No evidence of acute cardiovascular disease

Exclusion Criteria:

* Acute myocardial infarction in the last six months
* Pulmonary embolism in the last six months
* Hospitalisation for heart failure in the last six months
* Chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with clinically stable moderate aortic valve stenosis
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Cardiac troponin T | One year
Cardiac troponin I | One year
NT-pro-BNP | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Background] Klinkenberg LJ, van Dijk JW, Tan FE, van Loon LJ, van Dieijen-Visser MP, Meex SJ. Circulating cardiac troponin T exhibits a diurnal rhythm. J Am Coll Cardiol. 2014 May 6;63(17):1788-95. doi: 10.1016/j.jacc.2014.01.040. Epub 2014 Feb 26. PMID 24583293
- [Derived] Peeters FECM, Kietselaer BLJH, Hilderink J, van der Linden N, Niens M, Crijns HJGM, Meex SJR. Biological variation of cardiac markers in patients with aortic valve stenosis. Open Heart. 2019 May 8;6(1):e001040. doi: 10.1136/openhrt-2019-001040. eCollection 2019. PMID 31168392